CLINICAL TRIAL: NCT04318119
Title: Cerebral Small Vessel Disease Registry Study
Status: Recruiting | Type: Observational
Sponsor: Bin Cai (Other)
Responsible Party: Sponsor-Investigator, Bin Cai, Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2019]245
Record Dates: First submitted 2020-03-14; First posted 2020-03-23 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cerebral Small Vessel Diseases
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of Cerebral Small Vessel Disease (CSVD) and in a prospective multicenter study, to assess the clinical, genetic and epigenetic features of patients with CSVD, , to find independent imaging markers, and to optimize clinical management.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent.
2. Age>18
3. At least one of the following CSVD MRI characteristics: ①recent small subcortical infarct;②lacune of presumed vascular origin;③white matter hypertensity of presumed vascular origin;④perivascular space;⑤cerebral microbleeds;⑥brain atrophy

Exclusion Criteria:

1. Unable to cooperate with inspectors
2. Non-vascular white matter lesions
3. Other cognitive diseases (such as alzheimer's disease, Parkinson's disease or thyroid disease)
4. Serious systemic illness, such as heart, liver, kidney disease or major mental illness
5. Contraindications for imaging examination

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who are diagnosed as Cerebral Small Vessel Disease
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2049-11-18 (Estimated); Study Completion 2055-11-18 (Estimated)

PRIMARY OUTCOMES:
Overall outcomes in patients with cerebral small vessel disease. | From date of enrollment until the date of death from any cause, assessed up to 30 years
  record the occurrence of stroke and use modified Rankin Scale (mRS) to measure the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.

SECONDARY OUTCOMES:
the development of the burden of microbleeds in MRI | From date of enrollment until the date of death from any cause, assessed up to 30 years
  using MARS scale to evaluate the development of the burden of microbleeds
the development of the burden of white matter hypertension in MRI | From date of enrollment until the date of death from any cause, assessed up to 30 years
  using Fazakes scale to evaluate the development of the burden of white matter hypertension
the development of lacunes in MRI | From date of enrollment until the date of death from any cause, assessed up to 30 years
  record the number and location of lacunes
the development of enlarged perivascular space in MRI | From date of enrollment until the date of death from any cause, assessed up to 30 years
  record the number and location of enlarged perivascular space

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology , First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Hu F, Xie W, Fan M, Wang Y, Xu S, Qiu W, Yang T, Lv H, Huang H, Wu Y, Fu Y, Cai B. Intracerebral Hemorrhage in Autosomal Dominant Cerebral Arteriopathy With Subcortical Infarcts and Leukoencephalopathy. Eur J Neurol. 2025 Mar;32(3):e70100. doi: 10.1111/ene.70100. PMID 40067051